CLINICAL TRIAL: NCT03510338
Title: A Pharmacoscintigraphic Clinical Study to Evaluate a Biphasic Release Sildenafil Formulation (With Immediate and Sustained Release Components) Compared to a Marketed Sildenafil Product in Fed and Fasted States
Brief Title: Pharmacoscintigraphic Study to Evaluate Two Sildenafil Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: N4 Pharma UK Ltd. (Industry)
Collaborators: BDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BC230
Record Dates: First submitted 2018-04-12; First posted 2018-04-27 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sublingual sildenafil (fasted) (Experimental): Subjects receive a single dose of 100 mg sildenafil
  Interventions: Drug: Sublingual sildenafil
- Oral sildenafil (fed) (Active Comparator): Subjects receive a single dose of 50 mg sildenafil (Viagra)
  Interventions: Drug: Oral sildenafil
- Sublingual sildenafil (fed) (Experimental): Subjects receive a single dose of 100 mg sildenafil
  Interventions: Drug: Sublingual sildenafil
- Oral comparator (fasted) (Active Comparator): Subjects receive a single dose of 50 mg sildenafil (Viagra)
  Interventions: Drug: Oral sildenafil

INTERVENTIONS:
Drug: Sublingual sildenafil — 100 mg biphasic sildenafil tablet
  Other Names: N4S001
  Arms: Sublingual sildenafil (fasted); Sublingual sildenafil (fed)
Drug: Oral sildenafil — 50 mg oral sildenafil (Viagra)
  Other Names: Viagra
  Arms: Oral comparator (fasted); Oral sildenafil (fed)

SUMMARY:
The study will assess a new biphasic release sildenafil formulation (N4S001), developed by N4 Pharma. The N4S001 tablet contains a total of 100 mg sildenafil.

The N4S001 tablet is designed to provide a faster onset of release and a longer therapeutic window compared to currently marketed sildenafil products.

This is a single centre, open-label, four-arm crossover study in up to 12 healthy male volunteers.

The following treatments will be dosed:

Assessment Visit 1: N4S001 tablet containing 100 mg sildenafil (fasted)

Assessment Visit 2: N4S001 tablet containing 100 mg sildenafil (fed)

Assessment Visit 3: Viagra film-coated tablet containing 50 mg sildenafil (fasted)

Assessment Visit 4: Viagra film-coated tablet containing 50 mg sildenafil (fed)

The immediate release layer of each N4S001 tablet will be radiolabelled to contain 4 MBq (megabecquerel) 99mTc at time of dose.

DETAILED DESCRIPTION:
A pharmacoscintigraphic clinical study will be undertaken to quantify the scintigraphic kinetics and extent of dispersion of the immediate release portion of the N4S001 tablet in the oral cavity, and to measure sildenafil and its main metabolite, N-desmethyl sildenafil, in the blood plasma. The study will comprise an open-label, four-treatment crossover study in up to 12 healthy male volunteers. All subjects will receive four treatments throughout the study. The initial fast onset release portion of each N4S001 tablet will be radiolabelled to enable the dispersion characteristics of this part of the formulation to be investigated in-vivo. The immediate release portion of the N4S001 tablet will be radiolabelled to contain approximately 4 MBq technetium-99m (99mTc) at time of dose (TOD). Blood samples will be taken at pre-defined times to allow pharmacokinetic (PK) evaluation of drug absorption of the N4S001 tablet and of the reference product, Viagra 50 mg film coated tablets. Blood pressure will be recorded at set time intervals to assess the effects of the N4S001 tablet against the reference product. Subjects will also assess the taste acceptability of the N4S001 tablet using a 7-point categorical scale and oral examinations will be completed to assess any local oral effects of N4S001.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18 and 65 years inclusive
* BMI between 18 and 30 kg/m2 inclusive
* Body weight ≥50 kg
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any trial related activities
* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination

Exclusion Criteria:

* Current or recurrent disease that, in the opinion of the physician responsible, could affect the study conduct or laboratory assessments (e.g. hepatic disorders, renal insufficiency, congestive heart failure).
* Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
* A history of current or relevant previous non self-limiting gastrointestinal disorders.
* Currently suffering from disease known to impact gastric emptying, e.g. migraine, Type 1 or Type 2 diabetes mellitus.
* Currently suffering from any oromucosal condition (e.g. salivary gland disorders, xerostomia, aphthous ulcers) or recent oral surgery that in the opinion of the physician responsible could interfere with the study objectives.
* Currently or previously suffering from non-arteritic anterior ischaemic optic neuropathy (NAION).
* Known hereditary degenerative retinal disorders such as retinitis pigmentosa.
* Hypotension (blood pressure <90/50 mmHg).
* Recent history of stroke or myocardial infarction.
* Laboratory screening results that suggest an abnormal liver and/or renal function.
* Subject has a screening QTc value of greater than or equal to 450 msec or an ECG that is not suitable for QTc measurements (e.g. poorly defined termination of the T-wave). The ECG taken at screening must be considered not clinically significant by the Investigator/ study physician.
* As a result of a physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
* Subject has taken prescribed medication within 14 days prior to the first assessment visit which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety. Subjects will be withdrawn from subsequent study days if they commence taking prescribed medication during the study period which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety.
* Subject has taken over-the-counter (OTC) medication within 48 hours prior to the first assessment visit. This includes the use of vitamins and natural or herbal remedies. Subjects who have taken OTC medication may still be entered into the study if, in the opinion of the physician responsible, the medication will not interfere with the study procedures or compromise safety.
* Concomitant use of other phosphodiesterase 5 (PDE5) inhibitors, or other pulmonary arterial hypertension (PAH) treatments containing sildenafil (REVATIO), or other treatments for erectile dysfunction.
* Concomitant use of antihypertensive medications (e.g. diuretics, angiotensin converting enzyme (ACE) inhibitors etc).
* Concomitant use of nitrate medications.
* Recent history (within the last year) of alcohol or other substance abuse.
* Subject has an average weekly alcohol intake of greater than 21 units.
* Subject has positive urine drugs of abuse test at screening.
* Subject has a positive breath alcohol test at screening.
* Subject has recently discontinued smoking (less than 3 months).
* Subject is currently a smoker or user of nicotine-containing products.
* Subject has a positive urine cotinine test at screening.
* Subject has a history of allergy to sildenafil, to any component of the dosage form, or any other allergy, which in the opinion of the physician responsible, contraindicates their participation.
* Has an allergy to any of the contents of the standardised meals.
* Subject is vegetarian.
* Subject is lactose intolerant.
* Participation in another clinical study (inclusive of final post-study examination) or receipt of an investigational drug within the 12 weeks before first screening visit.
* Previous participation in this study.
* Subject whose participation in this study will result in participation in more than four studies over a twelve month period.
* An employee of the sponsor, client or study site or members of their immediate family.
* Subjects for whom participation in this study will exceed the limits of total radiation exposure allowed in the previous twelve month period (5 mSv), or will exceed 10 mSv over the previous three year period.
* Subjects who are intending to father a child in the 3 months following the study or are unwilling to abstain from sexual intercourse with pregnant or lactating women.
* Subjects who are unwilling to use a condom/spermicide in addition to having their female partner use another form of contraception such as an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the assessment visit until 3 months following the study.
* Subject has donated blood or experienced significant blood loss within 3 months of screening and for the duration of the study.
* Difficulty accessing forearm veins for cannulation or blood sampling.
* Subject has any non-removable metal objects such as metal plates, screws etc in their chest or abdominal area, which in the opinion of the investigator, could affect the study conduct.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male volunteers aged 18-65 years
Enrollment: 12 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Sildenafil plasma concentrations | 24 hours
  Measure sildenafil and its main metabolite in plasma and compare pharmacokinetic profiles with that of a marketed sildenafil product in fed and fasted states

SECONDARY OUTCOMES:
Extent of dispersion | 1 hour
  Quantification of extent of dispersion of the immediate release portion of the radiolabelled N4S001 tablet in the oral cavity using gamma scintigraphy
Visualisation of kinetics | 1 hour
  Quantification the kinetics in the oral cavity of the immediate release portion of the radiolabelled N4S001 tablet using gamma scintigraphy
Change in oral examination findings post-dose | 1 hour
  Assess changes in the oral cavity following dosing of the N4S001 tablet
Blood pressure | 24 hours
  Systolic & diastolic measurements will be used to assess the effects of the N4S001 tablet compared with the marketed sildenafil product
Heart Rate | 24 hours
  Measurements will be used to assess the effects of the N4S001 tablet compared with the marketed sildenafil product
Questionnaire | 1 hour
  Assessment of taste acceptability using a 7-point categorical scale

CONTACTS AND LOCATIONS:
Overall Officials: Howard NE Stevens, FRPharmS, Principal Investigator — BDD Pharma Ltd
Locations (1):
- BDD Pharma Ltd, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No